CLINICAL TRIAL: NCT04591483
Title: An Observational Prospective Natural History Study of Stargardt-like Macular Dystrophy (STDG3) Secondary to Mutations in ELOVL4
Brief Title: Stargardt-like Macular Dystrophy (STDG3) Secondary to Mutations in ELOVL4
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000108; 000108-EI
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09-30

CONDITIONS: Stargardt-Like Macular Dystrophy
Keywords: ABCA4; Oral Metformin; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected: Patients with Stargardt-like macular dystrophy 3 who are >= 10 years of age.

SUMMARY:
Background:

STDG3 is an inherited eye disease. Currently there is no treatment for STDG3. Past studies of STDG3 have largely looked at members of large families at a single time point. Researchers want to learn more about the disease at an individual level.

Objective:

To understand the natural history of changes in the retina that occur in people with STDG3.

Eligibility:

People ages 10 and older with STDG3 due to a variant in the ELOVL4 gene.

Design:

Participants will have 6 visits. First they will have a screening visit, followed by a baseline visit. Then they will have a visit 6 months later. Then they will have a visit 1, 2, and 3 years after the first visit. Visits will last 4 to 8 hours.

Visits will include the following:

Medical history and physical exam.

Complete eye exam. Participants' eye pressure and ability to see letters on a vision chart will be tested. Their pupils will be dilated with eye drops. Pictures will be taken of the retina and the inside of the eye.

Questions about participants' family history, especially the presence of eye disease.

Visual field test. Participants will be seated in front of a large dome and asked to press a button when they see a light within the dome.

Electroretinogram. Participants will sit in the dark with their eyes patched for 30 minutes. Then they will wear special contact lenses and watch flashing lights.

Optical coherence tomography. Cross-sectional pictures will be taken of participants' retinas.

Fundus autofluorescence. Blue light will be shone into participants eyes to assess the health of the retina....

DETAILED DESCRIPTION:
Title: An Observational Prospective Natural History Study of Stargardt-like Macular Dystrophy (STDG3) Secondary to Mutations in ELOVL4

Study Description: Potential therapeutics for Stargardt-like macular dystrophy (STDG3) have been proposed. Cross-sectional studies of large families suggest progressive macular atrophy in STDG3 but there is a paucity of longitudinal data for these patients. The overall goal is to establish a natural history study of STDG3.

Objectives: The primary objective is to assess the longitudinal changes in retinal structure in STDG3 patients.

The secondary objective is to assess the longitudinal changes in retinal function in STDG3 patients.

An exploratory objective is to assess the longitudinal changes in functional vision and the participant s perceived effect on activities of daily living (e.g., mobility).

Endpoints: The primary endpoints are: A) the growth rate of the square root area of loss of the inner segment/outer segment band (EZband) obtained from spectral-domain optical coherence tomography (SD-OCT) and B) the rate of atrophy enlargement obtained from fundus autofluorescence

The secondary endpoints are: A) the change in BCVA total letters read from baseline to Year 3 and B) the rate of loss of retinal sensitivity measured with perimetry

Study Population: Up to 25 patients with Stargardt-like macular dystrophy 3 who are >= 10 years of age.

Description of Sites/Facilities Enrolling Participants: Patients will be seen in the Ophthalmic Genetics Clinic at the National Eye Institute within the NIH Clinical Center in Bethesda.

Study Duration: 84 months (7 years).

Participant Duration: 36 months (3 years).

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Participant must be at least ten years of age.
3. Ability to perform required functional testing and ophthalmic imaging.
4. A mutation in ELOVL4 with a typical clinical presentation of Stargardt-like macular dystrophy.
5. Participant (or legal guardian) must understand and sign the protocol s informed consent document.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Two or more definitive mutations in ABCA4 and/or one mutation in RDS/peripherin or PROM1.
2. Systemic medical contraindications that are rarely associated with ELOVL4 (e.g., Spinocerebellar Ataxia-34).

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 25 patients with Stargardt-like macular dystrophy 3 who are >= 10 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2028-07-16 (Estimated); Study Completion 2028-07-16 (Estimated)

PRIMARY OUTCOMES:
Growth rate in square root area of loss of the inner segment/outer segment band (EZband) | Day 1, 182, 364, 728, 1,092
  The growth rate of the square root area of loss of the inner segment/outer segment band (EZband) obtained from SD-OCT.
Growth rate of square root area of atrophy measured from short-wavelength autofluorescence | Day 1, 182, 364, 728, 1,092
  The rate of atrophy enlargement obtained from fundus autofluorescence.

SECONDARY OUTCOMES:
The change in BCVA total letters read from baseline to Year 3 | Day 1, 182, 364, 728, 1,092
  The change in BCVA total letters read from baseline to Year 3.
The rate of loss of retinal sensitivity measured with perimetry | Day 1, 182, 364, 728, 1,092
  The rate of loss of retinal sensitivity measured with perimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Brett G Jeffrey, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000108-EI.html